CLINICAL TRIAL: NCT06851767
Title: Phase 1/2 Base-Edited Hematopoietic Stem/Progenitor Cell X-Linked Severe Combined Immunodeficiency Gene Therapy
Brief Title: Base-Edited Hematopoietic Stem/Progenitor Cell X-Linked Severe Combined Immunodeficiency Gene Therapy
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002273; 002273-I
Record Dates: First submitted 2025-02-26; First posted 2025-02-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11-14

CONDITIONS: X-linked Severe Combined Immunodeficiency; X-SCID; XSCID
Keywords: base editing; Gene Therapy
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases | interventions — plerixafor; Filgrastim; Fibroblast Growth Factor 7; Busulfan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental)
  Interventions: Genetic: Plerixafor; Drug: Filgrastim; Drug: Palifermin; Drug: Busulfan; Biological: Base-edited hematopoietic stem and progenitor cells

INTERVENTIONS:
Genetic: Plerixafor — Stem Cell Mobilizing Agent: Subcutaneous administration for 2 consecutive days to improve stem cell collection.
Drug: Filgrastim — Stem Cell Mobilizing Agent: Subcutaneous administration for 6 consecutive days. It is necessary to mobilize stem cells for collection.
Drug: Palifermin — Mucositis prophylaxis: As is standard practice prior to busulfan conditioning, IV infusion of keratinocyte growth factor (palifermin) will be administered at 60 micrograms/kg/day for 3 days before initiation of busulfan (days -6 to -4), as well as for the 3 days following study agent administration (days 1 to 3).
Drug: Busulfan — Transplant Conditioning Agent: An alkylating chemotherapy drug to enhance engraftment of the study agent (base-edited stem cells). For this study, busulfan is administered once daily (3 mg/kg) x 2 days, targeting a daily busulfan AUC of 4500-6500 micromol*min/L or a cumulative AUC of 9000 micromol*min/L (for the 2 days of therapy if levels are available. Busulfan will be infused over 3 hours each day as per standard clinical practice.
Biological: Base-edited hematopoietic stem and progenitor cells — Investigational/Study Agent: Base-edited autologous CD34 plus hematopoietic stem and progenitor cell product. A one-time dose >5(SqrRoot) 10^6 base-edited cells/kg body weight will be administered to each participant. The exact dosage depends on the number of viable cells that are repaired, cryopreserved, and thawed. The study agent will be administered by IV infusion in a volume of approximately 50 mL over about 15-30 minutes, in accordance with NIH CC DTM infusion policy.

SUMMARY:
Background:

X-linked severe combined immunodeficiency (XSCID) is a rare inherited disorder that affects the immune system. It is caused by a change in the IL2RG gene. Researchers are investigating a new type of gene therapy for people with XSCID. This technique, called base-edited stem cell transplants, involves collecting a person s own stem cells, editing the genes to repair IL2RG gene, and returning the edited cells to the person.

Objective:

To test base-edited stem cell transplants in people with XSCID.

Eligibility:

People aged 3 years and older with XSCID.

Design:

Participants will be screened. They will have a physical exam. They may give blood, urine, and stool samples. They may have tests of their heart and lung function. They may have fluid and cells drawn from their bone marrow.

Participants will undergo apheresis. Blood will be taken from the body through a needle inserted into 1 arm. The blood will pass through a machine that separates out the stem cells. The remaining blood will be returned to the body through a different needle. The collected stem cells will undergo gene editing.

Participants will be admitted to the hospital 1 week before treatment. They will receive a central line: A flexible tube will be inserted into a large vein. This tube will be used to administer drugs and draw blood during their stay. They will receive drugs to prepare their bodies for the treatment.

The base-edited stem cells will be infused through the central line. Participants will remain in the hospital for at least 3 weeks while they recover.

Follow-up visits will continue for 15 years.

DETAILED DESCRIPTION:
Study Description:

This is a phase 1/2, non-randomized study of a single infusion of autologous hematopoietic stem/progenitor cells base-edited to repair interleukin 2 receptor gamma (IL2RG) mutations (BE-HSPC IL2RG) in 18 participants with X-linked severe combined immunodeficiency (X-SCID).

Primary Objective:

Evaluate the safety of treatment with BE-HSPC IL2RG in participants with X-SCID.

Secondary Objectives:

Evaluate efficacy of treatment with BE-HSPC IL2RG in participants with X-SCID.

Exploratory Objectives:

1. Evaluate off-target (OT) editing activity.
2. Compare outcomes of immune reconstitution with lentivector (LV) gene therapy.

Primary Endpoint:

Safety of treatment with BE-HSPC IL2RG, by quantifying frequency and severity of adverse events (AEs) related to study agent from infusion to 12 months after infusion.

Secondary Endpoints (24 months post-study agent infusion):

1. Percentage of participants with >=5% mutation-repaired myeloid cells.
2. Editing efficiency in peripheral blood cells (such as T, B, and natural killer [NK] cells).
3. Immune reconstitution:

   1. T, B, and NK cell number improvement from baseline.
   2. Emergence of naive T cells and CD31+ recent thymic emigrants.
   3. B-cell function: immunoglobulin (Ig) production.
   4. Specific responses to vaccines.
4. Clinical efficacy: improvement from baseline problems such as recurrent infection, chronic norovirus, protein-losing enteropathy, gastrointestinal complaints, growth failure, malnutrition, or immune dysregulation.
5. Frequency and severity of all study agent-related AEs and serious adverse events (SAEs) from time of study product infusion.

Exploratory Endpoints:

1. Evaluate for frequency of off-targets (OTs) by high-throughput sequencing (HTS) of the target mutation at 2 years post-infusion.
2. Compare rates of immune reconstitution with LV-X-SCID gene therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged >= 3 years and weigh >=10 kg
* Patients with X-SCID
* If previously transplanted, must be >=18 months post-HSCT
* Expected survival of at least 120 days.
* Ability to undergo apheresis for stem cell collection.
* Patients with proven mutation in the common gamma chain gene as defined by direct sequencing of patient DNA. At this time, only patients with a IL2RG p.Q144X, IL2RG p.R289X, IL2RG p.Q235X and IL2RG p.R226H mutations can be treated.
* Participants of reproductive potential must agree to consistently use highly effective contraception throughout study participation and for at least 2 years post-treatment.

Acceptable forms of contraception are:

--For males: Condoms or other contraception with partner.

* Documented to be negative for HIV infection by PCR
* The patient must be judged by the primary evaluating physician to have a suitable family and social situation consistent with ability to comply with protocol procedures and the long-term follow-up requirements.
* Medical lab data (historical) of severe B cell dysfunction (low or absent IgG levels, failed immune response to vaccines);

OR

demonstrated requirement for intravenous gamma globulin (IVIG) (significant drop over 3 to 6 weeks between peak and trough IgG levels).

-Must be willing to have blood and tissue samples stored IN ADDITION, patients must satisfy the following Laboratory Criteria AND Clinical Criteria

Laboratory Criteria: (>=1 must be present)

* CD4+ lymphocytes: absolute number <= 50% of the lower limit of normal (LLN)
* CD4+CD45RA+ lymphocytes: absolute number <= 50% of the LLN OR T-cell receptor excision circles (TRECs) <= 5% of normal for age.
* Memory B Cells: absolute number <= 50% of LLN
* Serum IgM<normal for age
* NK cells: absolute number <= 50% of LLN
* Lymphocyte proliferative response to each of 2 mitogens, phytohemagglutinin (PHA) and concanavalin A (ConA), is <= 25% compared with a normal control.
* Molecular spectratype analysis- absent or very oligoclonal (1-3 dominant peaks) in >=6 of the 24 V(Beta) T-cell receptor families.

Clinical Criteria: (>=1 must be present)

I. Infections (not including molluscum, warts or mucocutaneous candidiasis; see VII and VIII below):

Three significant new or chronic active infections during the 2 years preceding evaluation for enrollment, with each infection accounting for one criterion.

Infections are defined as an objective sign of infection

* (fever >=38.3 degrees Celsius (101 degrees Fahrenheit) or
* neutrophilia or
* pain/redness/swelling or
* radiologic/ultrasound imaging evidence or
* typical lesion or histology or
* new severe diarrhea or
* cough with sputum production.

In addition to one or more of these signs/symptoms of possible infection, there also must be at least 1 of the following criteria as evidence of the attending physician s intent to treat a significant infection (a. and b.) or objective evidence for a specific pathogen causing the infection (c.)

1. Treatment (not prophylaxis) with systemic antibacterial, antifungal or antiviral antibiotics >=14 days

   OR
2. Hospitalization of any duration for infection

   OR
3. Isolation of a bacteria, fungus, or virus from biopsy, skin lesion, blood, nasal washing, bronchoscopy, cerebrospinal fluid or stool likely to be an etiologic agent of infection

II. Chronic pulmonary disease as defined by:

1. Bronchiectasis by x-ray computerized tomography

   OR
2. Pulmonary function test (PFT) evidence for restrictive or obstructive disease that is 60% of Predicted for Age

   OR
3. Pulse oximetry <=94% in room air (if patient is too young to comply with performance of PFTs).

III. Gastrointestinal enteropathy:

1. Diarrhea-watery stools >=3 times per day (of at least 3 months duration that is not a result of infection as defined in criterion I. above)

   OR
2. Endoscopic evidence (gross and histologic) for enteropathy (endoscopy will only be performed if medically indicated)

   OR
3. Other evidence of enteropathy or bacterial overgrowth syndrome: including malabsorption of fat soluble vitamin(s), abnormal D-xylose absorption, abnormal hydrogen breath test, evidence of protein losing enteropathy (for example increasingly high or frequent dosing of intravenous gamma globulin supplement required to maintain blood IgG level).

IV. Poor nutrition: Requires G-tube or intravenous feeding supplement to maintain weight or nutrition.

V. Auto- or allo-immunity: Examples must include objective physical findings that include, but are not limited to any one of alopecia, severe rashes at more than one anatomic site and not due to infection, uveitis, joint pain with redness or swelling or limitation of movement that is not a result of infection, lupus-like lesions, and granulomas (Does not include auto- or allo-immune enteropathy which is criterion iii). Where possible and appropriate, diagnosis will be supported by histopathology or other diagnostic modality.

VI. Failure to grow in height: <=3rd percentile for age

VII. Skin molluscum contagiosum OR warts (this criterion is satisfied if molluscum consists of >=10 lesions or there are two or more lesions at each of two or more widely separated anatomic sites; or there are >=3 warts at different anatomic sites at the same time; or the patient has both molluscum and warts)

VIII. Mucocutaneous candidiasis (chronic oral thrush or candida esophagitis or candida intertriginous infection or candida nail infections; must be culture positive to satisfy this criterion)

IX. Hypogammaglobulinemia: requires regular IgG supplementation

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Available HLA-matched sibling donors.
* Known hypersensitivity to busulfan or any component of the product.
* Contraindications for administration of busulfan.
* Childhood malignancy (occurring before 18 years of age) in the participant or a first degree relative, or previously diagnosed known genotype of the participant conferring a predisposition to cancer unless approved by the Hematology consult team (no DNA or other testing for cancer predisposition genes will be performed as part of the screen for this protocol).
* Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the participant, or would preclude the patient from successful study completion.

Ages: 3 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantify frequency and severity of adverse events (AEs) related to study agent from infusion to 12 months after infusion. | 12 months
  Evaluate the safety of treatment with BE-HSPC IL2RG in participants with X-SCID.

SECONDARY OUTCOMES:
Evaluate percentage of participants with >= 5% mutation-repaired alleles in PBMCs. | 24 months
  Measure efficacy of treatment by assessing efficiency of base editor at repair of mutations.
Evaluate editing efficiency in peripheral blood cells (such as T, B, and natural killer [NK] cells). | 24 months
  Measure efficacy of treatment by assessing molecular evidence for mutation repair.
Evaluate Immune reconstitution: a. T, B, and NK cell number improvement from baseline. b. Emergence of naive T cells and CD31+ recent thymic emigrants.c. B-cell function: immunoglobulin (Ig) production. d. Specific responses to vacci... | 24 months
  Measure efficacy of treatment by assessing immune reconstitution as indicated by 1) increase in immune cell numbers; 2) restoration of thymic function with production of na(SqrRoot) ve T cells and CD31+ T cells; 3) Evaluate restoration of B-cell function.
Evaluate clinical efficacy by improvement from baseline problems such as recurrent infection, chronic norovirus, protein-losing enteropathy, gastrointestinal complaints, growth failure, malnutrition, or immune dysregulation. | 24 months
  Measure efficacy of treatment by assessing comparison of clinical status before and after treatment as indicator of response to improved immune function.
Evaluate frequency and severity of all study agent-related AEs and serious adverse events (SAEs) from time of study product infusion. | 24 months
  Measure efficacy of treatment by assessing intervention-related AE rate.

CONTACTS AND LOCATIONS:
Overall Officials: Suk S De Ravin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002273-I.html